CLINICAL TRIAL: NCT07048678
Title: Evaluating the Impact of Preoperative Respiratory Exercises on Post-Surgical Pulmonary Outcomes: A Randomized Controlled Trial
Brief Title: Evaluating the Impact of Preoperative Respiratory Exercises on Post-Surgical Pulmonary Outcomes RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSAHSW/Batch-Fall23/907
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases | interventions — Standard of Care; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preoperative respiratory exercises (Experimental)
  Interventions: Combination Product: preoperative respiratory exercises
- Standard Care (Control Group) (Active Comparator)
  Interventions: Combination Product: Standard Care (Control Group)

INTERVENTIONS:
Combination Product: preoperative respiratory exercises — Participants in Group 1 will receive a combination of preoperative respiratory exercises designed to improve lung function and reduce the risk of postoperative pulmonary complications. The intervention includes:
  Arms: preoperative respiratory exercises
Combination Product: Standard Care (Control Group) — Participants in Group 2 will receive standard preoperative care provided by the hospital, which includes routine instructions related to surgery such as fasting guidelines, medication administration, and anesthesia protocols. No preoperative respiratory exercises (incentive spirometry, chest physiotherapy, or deep breathing exercises) will be provided to this group. This group serves as a control to compare the outcomes with the intervention group.
  Arms: Standard Care (Control Group)

SUMMARY:
This randomized controlled trial aims to evaluate the role of preoperative respiratory exercises in reducing postoperative pulmonary complications (PPCs) such as atelectasis, pneumonia, and hypoxia, and in shortening the hospital stay in surgical patients. A total of 126 adult patients (>40 years), scheduled for total knee or hip replacement surgeries at Horizon Hospital Lahore, will be randomly assigned into two groups: the intervention group and the control group.

DETAILED DESCRIPTION:
The intervention group will receive preoperative respiratory exercises including incentive spirometry, deep breathing exercises, and chest physiotherapy, one day before surgery. The control group will receive standard preoperative care without any respiratory exercises. Clinical assessments post-surgery will determine the presence of PPCs and hospital stay duration.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged over 40 years.
* Scheduled for total knee replacement (TKR) or total hip replacement (THR) surgery.
* Able to understand and follow instructions (cognitively intact).
* Provide informed consent to participate.

Exclusion Criteria:

* Patients will be excluded from the study if they meet any of the following conditions:
* Age below 40 years.
* Pregnancy.
* Edentulous patients (patients with no teeth).
* Patients with spinal or backbone injuries.
* Patients with contraindications to incentive spirometry or chest physiotherapy (e.g., recent eye surgery, rib fractures).
* Patients with impaired cognitive function who are unable to perform respiratory exercises correctly.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pulmonary Complication (PPC) assessment | 12 Months
  Postoperative Pulmonary Complication (PPC) assessment involves evaluating various risk factors to predict the likelihood of respiratory complications after surgery. The ARISCAT score is a widely used tool for this purpose, assigning points based on factors like age, preoperative oxygen saturation, respiratory infection history, anemia, surgical incision type, surgery duration, and whether it was an emergency procedure. Other assessment methods include the PPC Risk Prediction Score (focused on lung function, weight loss, and incision type) and indices like the Shapiro index and PI score

CONTACTS AND LOCATIONS:
Locations (1):
- Horizon hospital, 03, 404, 436 Block D-II, M.A Block D 2, Phase 1, Johar Town, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No